CLINICAL TRIAL: NCT00715767
Title: Correlation of Cognitive and Technical Skills Assessment for Basic Life Support and Identification of Barriers to Cross-Cultural Education
Brief Title: Basic Life Support (BLS) and Barriers to Cross-Cultural Education
Acronym: BLSinBotswana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Laerdal Medical (Industry)
Responsible Party: Pete Meaney, MD, Children's Hospital of Philadelphia
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 2008-1-5700
Record Dates: First submitted 2008-07-14; First posted 2008-07-15 (Estimated); Last update posted 2010-10-14 (Estimated); Status verified 2010-10

CONDITIONS: Medical Education
Keywords: BLS training; CPR; post graduate education; resource-limited settings; medical education; CPR retention; cultural barriers
MeSH Terms: interventions — Restraint, Physical; Mental Status and Dementia Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Assessment — Cognitive Assessment:
  Knowledge base and critical thinking will be evaluated by a 50-question BLS multiple-choice examination. At the designated 4 cognitive assessments in the study (pre-course, immediately post course, 3 months and 6 months) 50 equivalent questions will be used to cover all core BLS objectives. Technical Skills Assessment:
  Primary outcome measures of adequacy of chest compressions and ventilations as well as key actions for each of the 3standardized basic life support skill tests during 3-minute testing scenarios. Video review by 2independent experts will be utilized for objective assessment of time and order dependent skills, and manikin output will be utilized to assess qualitative effectiveness of skills (adequate ventilation, compression, and defibrillation).
  Survey Instrument for Barriers to Acute Medicine Education:
  A survey tool will be used to identify barriers to acute medicine education implementation and efficacy.
  Other Names: cognitive assessment; critical thinking; outcome measures of adequacy of chest compressions; outcome measures of adequacy of ventilations

SUMMARY:
This is a randomized, multi-center intervention trial comparing two educational programs on healthcare provider performance in the Botswana national hospital system. This study addresses the critical question of how to effectively and consistently measure and associate CPR knowledge and psychomotor skills, enabling the optimization of the learners' environment.

DETAILED DESCRIPTION:
Context: The World Health Organization (WHO) estimates that more than 16 million people die from cardiovascular diseases each year, accounting for more than one-third of global deaths. Almost half of these deaths take place in hospitalized settings. Standard acute medicine education programs have had limited success in training hospital based healthcare providers to acquire, retain, and transfer knowledge and skills to impact patient outcomes in both developed and developing countries. There is a gap between the cognitive knowledge and critical thinking skills attained during courses and the technical and team skills actually performed by hospital-based healthcare providers. This gap between existing knowledge and performed skills restricts care delivery, underutilizes available resources, and contributes to the number of preventable deaths. This gap is further accentuated in resource limited settings, where barriers to implementation of successful acute medicine training programs are often accentuated.

Primary Objective:

1. To determine selected cognitive knowledge and critical thinking skills which are associated with technical and team skills performance assessed immediately following Basic Life Support (BLS) for Health Care Providers course training.

Secondary Objectives:

1. To identify cultural, healthcare environment and educational barriers that currently impede acquisition, retention, and transfer of knowledge and skills in acute medicine educational programs in resource limited settings.

ELIGIBILITY:
Inclusion Criteria:

1. Healthcare providers involved in patient contact.
2. Participation in BLS for Healthcare Provider Course

Exclusion Criteria:

1. Have received formal Basic Life Support training in previous 12 months.
2. Inability to perform or complete cognitive and skills assessment testing (pre, immediate post, 3 or six month post).
3. Healthcare personnel performing an educational rotation at the district or referral hospital will not be eligible due to loss of follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2009-01; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To determine selected cognitive knowledge and critical thinking skills. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pete Meaney, MD, Principal Investigator — Children's Hospital of Philadelphia